CLINICAL TRIAL: NCT03976986
Title: Assessment of Portable Oxygen Concentrators in Infants Undergoing Hypoxic Challenge Testing. A Randomized Crossover Study.
Brief Title: Assessment of Portable Oxygen Concentrators in Infants Undergoing Hypoxic Challenge Testing.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Son Espases (Other)
Responsible Party: Principal Investigator, Sebastian Sailer, Principal Investigator, Hospital Son Espases
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: cop2016
Record Dates: First submitted 2019-05-31; First posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Hypoxia, Altitude
Keywords: Infants; Hypoxia Altitude Simulation Test; Oxygen Delivery Device; Portable Oxygen Concentrator; Hypoxic Challenge Testing
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cPOC - pPOC (Experimental): Randomized crossover study (according to a random number table): Patients are allocated randomly to two study groups (cPOC/pPOC). In case of Sat.O2 drop ≤ 85% during HCT, oxygen is administered by cPOC (continuous-flow). For patients who show a positive POC hypoxic reversal, HCT is repeated at 24 hours and oxygen is administered by pPOC (pulsed-flow).
  Interventions: Device: continuous-flow portable oxygen concentrator (cPOC); Device: pulsed-flow portable oxygen concentrator (pPOC)
- pPOC - cPOC (Experimental): Randomized crossover study (according to a random number table): Patients are allocated randomly to two study groups (cPOC/pPOC). In case of Sat.O2 drop ≤ 85% during HCT, oxygen is administered by pPOC (pulsed-flow). For patients who show a positive POC hypoxic reversal, HCT is repeated at 24 hours and oxygen is administered by cPOC (continuous-flow).
  Interventions: Device: continuous-flow portable oxygen concentrator (cPOC); Device: pulsed-flow portable oxygen concentrator (pPOC)

INTERVENTIONS:
Device: continuous-flow portable oxygen concentrator (cPOC) — SeQal Eclipse 3® on continuous-flow (SeQual,Ball Ground,GA): flow rate 2 litre per minute (lpm).
Device: pulsed-flow portable oxygen concentrator (pPOC) — InogenOne G3® (Inogen,Goleta,CA) on pulsed-flow mode: setting 2 (flow rate 420 ml/min, 16.8 ml +/- 3ml per bolus at 25 rpm).

SUMMARY:
Hypoxic Challenge Testing (HCT) is the recommended method for inflight hypoxia risk assessment. Onboard oxygen administration remains controversial. The Federal Aviation Administration approved portable oxygen concentrators (POCs) for onboard oxygen supply but there is lack of evidence about the use, especially in children. The aim of our study is to establish the effectiveness and safety of POCs in infants undergoing HCT.

DETAILED DESCRIPTION:
According to a forecast by International Air Transport Association the number of people travelling on commercial aircrafts is predicted to rise up to 8.2 billion passengers in 2037. Therefore evidence-based flight recommendations will gain importance in the future, especially for patients suffering from chronic diseases. Hypoxic Challenge Testing (HCT) is the recommended method for inflight hypoxia risk assessment where nitrogen is introduced in a plethysmograph reducing FiO2 (fraction of inspired oxygen) to 0.15. Oxygen supply is recommended if PaO2 (partial pressure of oxygen in arterial blood) drops <50-55 mmHg (in adults) or Sat.O2 (oxygen saturation) ≤ 85% (in infants) where non-invasive pulse oximetry is the recommended method for hypoxia assessment. Onboard oxygen administration remains controversial. The effectiveness of pulsed-dosed systems remains unclear in small patients due to shallow breathing patterns. The aim of our study is to establish the effectiveness and safety of POCs in infants undergoing HCT.

ELIGIBILITY:
Inclusion Criteria:

Patients with baseline Sat.O2 >94% AND

* <1 year with neonatal respiratory disease
* required oxygen supply in the last 6 months
* chronic respiratory disease (eg cystic fibrosis, obstructive or restrictive pulmonary disease) with FEV 1 (forced expiratory volume in 1 second) or FVC (forced vital capacity) <50%.

Exclusion Criteria:

* acute respiratory infection

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2016-02-11 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

PRIMARY OUTCOMES:
Assessment of portable oxygen concentrators (POCs) to change HCT induced hypoxia (Sat.O2 drop ≤ 85%). | 20 minutes
  Hypoxia (Sat.O2 drop ≤ 85%) measured by Masimo SET Radical-7 Electron® pulse oximeter is induced performing HCT. Thereafter oxygen is administered through cPOC or pPOC until baseline Sat.O2 (Sat.O2 >93%) is achieved.

SECONDARY OUTCOMES:
POC comparison to change HCT induced hypoxia (Sat.O2 drop ≤ 85%). | 20 minutes
  Compare the capacity of different POCs: continuous flow (cPOC) versus pulsed flow (pPOC) to change HCT induced hypoxia (Sat.O2 ≤ 85%) until baseline Sat.O2 (Sat.O2 >93%) is achieved.
Relate patient age (months) to POCs capacity to change HCT induced hypoxia (Sat.O2 drop ≤ 85%). | 20 minutes
  Relationship between patient age (months) and POCs capacity to change hypoxic state (≤ 85%) to baseline Sat.O2 (>93%) measured by Masimo SET Radical-7 Electron®
Relate patient weight (kilograms) to POCs capacity to change HCT induced hypoxia (Sat.O2 drop ≤ 85%). | 20 minutes
  Relationship between patient weight (kilograms) and POCs capacity to change hypoxic state (≤ 85%) to baseline Sat.O2 (>93%) measured by Masimo SET Radical-7 Electron®

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Sailer, MD, Principal Investigator — Hospital Son Espases
Locations (1):
- Hospital Son Espases, Palma Mallorca, Mallorca, Spain

REFERENCES:
- [Result] Ahmedzai S, Balfour-Lynn IM, Bewick T, Buchdahl R, Coker RK, Cummin AR, Gradwell DP, Howard L, Innes JA, Johnson AO, Lim E, Lim WS, McKinlay KP, Partridge MR, Popplestone M, Pozniak A, Robson A, Shovlin CL, Shrikrishna D, Simonds A, Tait P, Thomas M; British Thoracic Society Standards of Care Committee. Managing passengers with stable respiratory disease planning air travel: British Thoracic Society recommendations. Thorax. 2011 Sep;66 Suppl 1:i1-30. doi: 10.1136/thoraxjnl-2011-200295. No abstract available. PMID 21856702
- [Result] Gong H Jr, Tashkin DP, Lee EY, Simmons MS. Hypoxia-altitude simulation test. Evaluation of patients with chronic airway obstruction. Am Rev Respir Dis. 1984 Dec;130(6):980-6. doi: 10.1164/arrd.1984.130.6.980. PMID 6508019
- [Result] Blakeman TC, Rodriquez D Jr, Gerlach TW, Dorlac WC, Johannigman JA, Branson RD. Oxygen requirement to reverse altitude-induced hypoxemia with continuous flow and pulsed dose oxygen. Aerosp Med Hum Perform. 2015 Apr;86(4):351-6. doi: 10.3357/AMHP.4184.2015. PMID 25945551
- [Result] Fischer R, Wanka ER, Einhaeupl F, Voll K, Schiffl H, Lang SM, Gruss M, Ferrari U. Comparison of portable oxygen concentrators in a simulated airplane environment. Respir Med. 2013 Jan;107(1):147-9. doi: 10.1016/j.rmed.2012.10.001. Epub 2012 Oct 22. PMID 23085214
- [Result] Bunel V, Shoukri A, Choin F, Roblin S, Smith C, Similowski T, Morelot-Panzini C, Gonzalez J. Bench Evaluation of Four Portable Oxygen Concentrators Under Different Conditions Representing Altitudes of 2438, 4200, and 8000 m. High Alt Med Biol. 2016 Dec;17(4):370-374. doi: 10.1089/ham.2016.0056. PMID 27959667
- [Result] Chen JZ, Katz IM, Pichelin M, Zhu K, Caillibotte G, Finlay WH, Martin AR. In Vitro-In Silico Comparison of Pulsed Oxygen Delivery From Portable Oxygen Concentrators Versus Continuous Flow Oxygen Delivery. Respir Care. 2019 Feb;64(2):117-129. doi: 10.4187/respcare.06359. Epub 2019 Jan 29. PMID 30696754